CLINICAL TRIAL: NCT04568421
Title: Argentinian Registry of Patients With Rheumatic Diseases and COVID-19 Infection
Acronym: SAR-COVID
Status: Completed | Type: Observational
Sponsor: Sociedad Argentina de Reumatologia (Other)
Responsible Party: Sponsor
Other Study IDs: 01
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Rheumatic Diseases
Keywords: COVID-19
MeSH Terms: conditions — Rheumatic Diseases; COVID-19 | interventions — Immunosuppressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treated with immunomodulatory and/or -suppressive drugs: Patients with rheumatic diseases treated with immunomodulatory and/or immunosuppressive drugs and with diagnosis of SARS-CoV-2 infection (past or present) with positive test for the virus SARS-CoV-2 from analysis of nasopharyngeal or oropharyngeal swab specimens (reverse transcriptase-polymerase- chain-reaction assay) or by serology, independently of symptoms.
  Interventions: Drug: Immunosuppressive Agents
- Not treated with immunomodulatory and/or -suppressive drugs: Patients with rheumatic diseases not treated with immunomodulatory and/or immunosuppressive drugs and with diagnosis of SARS-CoV-2 infection (past or present) with positive test for the virus SARS-CoV-2 from analysis of nasopharyngeal or oropharyngeal swab specimens (reverse transcriptase-polymerase- chain-reaction assay) or by serology, independently of symptoms.

INTERVENTIONS:
Drug: Immunosuppressive Agents — Immunomodulatory and/or immunosuppressive drugs according to the indication of the treating physician
  Other Names: Immunomodulatory and/or immunosuppressive treatments
  Groups: Treated with immunomodulatory and/or -suppressive drugs

SUMMARY:
SAR-COVID is a national, multicenter, prospective, observational longitudinal registry of consecutive patients with diagnosis of rheumatic diseases treated or not with immunomodulatory and/or immunosuppressive drugs and SARS-CoV-2 infection (asymptomatic or COVID-19).

Hypothesis: Patients with rheumatic diseases who are under chronic treatment with immunomodulatory and/or immunosuppressive drugs more frequently have an asymptomatic infection, a milder COVID-19 and lower mortality than patients with rheumatic diseases without immunomodulatory and/or immunosuppressive treatments.

DETAILED DESCRIPTION:
SAR-COVID is a national, multicenter, prospective, observational longitudinal registry of consecutive patients with diagnosis of rheumatic diseases treated or not with immunomodulatory and/or immunosuppressive drugs and SARS-CoV-2 infection (asymptomatic or COVID-19).

HYPOTESIS: Patients with rheumatic diseases who are under chronic treatment with immunomodulatory and/or immunosuppressive drugs more frequently have an asymptomatic infection, a milder COVID-19 and lower mortality than patients with rheumatic diseases without immunomodulatory and/or immunosuppressive treatments.

TARGET POPULATION: Patients > 18 years of age with any rheumatic disease. ELIGIBILITY CRITERIA Inclusion Criteria

* Age > 18 years.
* Patients with diagnosis of rheumatic diseases (treated or not with immunomodulatory and/or immunosuppressive drugs).
* Patients with diagnosis of SARS-CoV-2 infection (past or present) with positive test for the virus SARS-CoV-2 from analysis of nasopharyngeal or oropharyngeal swab specimens (reverse transcriptase-polymerase- chain-reaction assay) or by serology, independently of symptoms.

Exclusion Criteria

• Patients who do not wish to participate or are unable to give informed consent.

RECRUITMENT: All rheumatologists, members of the Argentine Society of Rheumatology will be invited to participate in the registry. It is expected that 3,000 patients with COVID-19 and some rheumatic disease, who are cared for by rheumatologists in any of the 23 provinces of Argentina, will be enrolled in the SAR-COVID registry during the period from July 1 to December 31, 2020. Twelve-month extension of the recruitment period will be applied if the expected number of patients is not achieved by the end of the inclusion date. Two cohorts will be included: the first will enroll 1,500 patients treated with immunomodulatory and/or immunosuppressive drugs, and the second will enroll 1,500 patients without immunomodulatory and/or immunosuppressive drugs.

DATA COLLECTION: All variables will be collected by self-report, clinical and laboratory examination and/or medical records review, performed by the rheumatologist during patient hospitalization due to COVID-19, or at the patient control visit performed after SARS-CoV-2 infection. The data will be entered into the ARTHROS eCRF (online application designed ad hoc), which in turn will facilitate generating queries and perform the statistical analysis.

PERIODIC REPORTS: Patients will be followed up for 12 months, in order to evaluate their evolution and identify the effect of the SARS-CoV-2 infection on their rheumatological disease. For this reason, in this registry the data will be collected in two phases:

* PHASE I: Corresponds to the baseline visit (T0). Sociodemographic data, diagnosis, symptoms, treatment, hospitalization, complications, characteristics of the rheumatic disease and its treatment before and during the infectious process will be recorded.
* PHASE II: This second visit (T1) will be carried out 12 months after patients registration. Its objective is to identify long-term complications after SARS-CoV-2 infection and to assess the impact of infection on rheumatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or older than 18 years.
* Patients with diagnosis of rheumatic diseases (treated or not with immunomodulatory and/or immunosuppressive drugs).
* Patients with diagnosis of SARS-CoV-2 infection (past or present) with positive test for the virus SARS-CoV-2 from analysis of nasopharyngeal or oropharyngeal swab specimens (reverse transcriptase-polymerase- chain-reaction assay) or by serology, independently of symptoms.

Exclusion Criteria:

* Patients who do not wish to participate or are unable to give informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19 and some rheumatic disease, who are cared for by rheumatologists in any of the 23 provinces of Argentina
Sampling Method: Non-Probability Sample
Enrollment: 2982 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 2 month
  Death caused by SARS-CoV-2 infection
Hospitalization | 2 month
  Hospitalization because of SARS-CoV-2 infection

SECONDARY OUTCOMES:
SARS-CoV-2 infection presentation | 1 month
  To describe clinical presentation of SARS-CoV-2 infection in patients with rheumatic diseases
Admission at the intensive care unit | 2 month
  Proportion of patients admitted at the intensive care unit
Invasive mechanical ventilation | 2 month
  Proportion of patients who required invasive mechanical ventilation
COVID-19 Complications | 2 month
  Proportion of patients who had complications associated with COVID-19 infection and describe them
Recovery rate | 2 month
  Proportion of patients fully or partially recovered after COVID-19 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Pons-Estel, Study Director — Unidad de Investigación Sociedad Argentina Reumatología
Locations (1):
- Sociedad Argentina de Reumatología, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isnardi CA, Soriano ER, Graf C, de la Vega MC, Pons-Estel BA, Roberts K, Quintana R, Gomez G, Yazdany J, Saurit V, Baez RM, Coello VVC, Pisoni CN, Berbotto G, Vivero F, Zelaya MD, Haye Salinas MJ, Reyes Torres AA, Ornella S, Nieto RE, Maldonado FN, Gamba MJ, Severina MLA, Tissera Y, Alba P, Cogo AK, Alle G, Gobbi C, Banos A, Velozo E, Pera M, Tanten R, Albiero JA, Maldonado Ficco H, Martire MV, Elkin MSG, Cosatti M, Cusa MA, Pereira D, Savio VG, Pons-Estel GJ. Does the Use of Immunosuppressive Drugs Impact on SARS-CoV-2 Infection Outcome? Data From A National Cohort of Patients With Immune-Mediated Inflammatory Diseases (SAR-COVID Registry). J Clin Rheumatol. 2023 Mar 1;29(2):68-77. doi: 10.1097/RHU.0000000000001903. Epub 2022 Nov 30. PMID 36454054
- [Derived] Isnardi CA, Roberts K, Saurit V, Petkovic I, Baez RM, Quintana R, Tissera Y, Ornella S, D Angelo Exeni ME, Pisoni CN, Castro Coello VV, Berbotto G, Haye Salinas MJ, Velozo E, Reyes Torres AA, Tanten R, Zelaya MD, Gobbi C, Alonso CG, de Los Angeles Severina M, Vivero F, Paula A, Cogo AK, Alle G, Pera M, Nieto RE, Cosatti M, Asnal C, Pereira D, Albiero JA, Savio VG, Maldonado FN, Gamba MJ, German NF, Banos A, Gallino Yanzi J, Galvez Elkin MS, Morbiducci JS, Martire MV, Maldonado Ficco H, Schmid MM, Villafane Torres JA, de Los Angeles Correa M, Medina MA, Cusa MA, Scafati J, Aguero SE, Lloves Schenone NM, Soriano ER, Graf C, Pons-Estel BA, Gomez G, Landi M, De la Vega MC, Pons-Estel GJ; S. A. R.-COVID Registry Investigators. Sociodemographic and clinical factors associated with poor COVID-19 outcomes in patients with rheumatic diseases: data from the SAR-COVID Registry. Clin Rheumatol. 2023 Feb;42(2):563-578. doi: 10.1007/s10067-022-06393-8. Epub 2022 Oct 6. PMID 36201124

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT04568421/Prot_SAP_000.pdf